CLINICAL TRIAL: NCT01526330
Title: A Double-blind, Randomized, Parallel, Placebo Controlled, Phase I/II Clinical Trial to Investigate the Safety, Tolerability and Efficacy of YH14618 Following Single Intradiscal Injection in Patients With Degenerative Disc Disease
Brief Title: Safety, Tolerability and Efficacy of YH14618 in Patients With Degenerative Disc Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YH14618-201
Record Dates: First submitted 2012-01-31; First posted 2012-02-03 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2014-07

CONDITIONS: Degenerative Disc Disease
Keywords: Degenerative disc disease; YH14618; Penial 2000; Penial 2K
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A (Experimental)
  Interventions: Drug: YH14618
- Group B (Experimental)
  Interventions: Drug: YH14618
- Group C (Experimental)
  Interventions: Drug: YH14618
- Group D (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YH14618 — A mg/disc
  Arms: Group A
Drug: YH14618 — B mg/disc
  Arms: Group B
Drug: YH14618 — C mg/disc
  Arms: Group C
Drug: Placebo — 0mg/disc
  Arms: Group D

SUMMARY:
The objective of this study is to assess the safety and tolerability of YH14618 during 24 weeks of follow-up period after single administration in patients with degenerative disc disease.

ELIGIBILITY:
Inclusion Criteria:

* Have signed a written informed consent voluntarily, prior to the any procedure
* Degenerative disc disease patients of aged over 20 years
* Have one or more of the symptomatic lumbar level(L1~S1) as confirmed using radiology(X-ray, MRI and/or discogram/CT)
* Have been diagnosed 2~3 degree of MRI index by modified thompson classification
* Oswestry diability index(ODI) of 30 or greater
* Visual analog scale(VAS) of 4 or greater

Exclusion Criteria:

* Subjects unable to have radiological examination
* Have history of neurological disease, herniated lumbar disc, compression fractures and lumbar spinal surgery
* Sacroiliac joint dysfunction
* Have been treated with any drugs for pain control within 7 days prior to the first administration
* Hypersensitivity to drugs
* Pregnant women, nursing mothers or subjects who do not agree to assigned contraception in the study
* Participated in any other clinical trials within 30 days prior to the first administration

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-05; Primary Completion 2014-01 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Evaulate the safety and tolerability after single intradiscal administation | 12 weeks of observational period
  Safety outcomes
  * Adverse events
  * 12-lead EKG
  * Physical examination
  * Standard lab results(hematology, blood chemistry, coagulation, urinalysis etc.)

SECONDARY OUTCOMES:
Change from baseline in disc height index at 12 week | Baseline, Week 12
Change from baseline in magnetic resonance imaging(MRI) index | Baseline, Week 12
Change from oswestry diability index(ODI) at week 12 | Baseline, Week 12
Change from baseline in visual analogue scale(VAS) at week 12 | Baseline, Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Young-joon Kwon, MD, PhD., Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- Kangbuk Samsung Medical Center, Seoul, South Korea